CLINICAL TRIAL: NCT06504953
Title: Evaluation of Anterior Tibial Knee Translation in Healthy Women With and Without Hormone Therapy
Acronym: LAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-PP-17
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Women; Tibial Translation; Hormone
Keywords: hormonale; anterior tibial translation; knee; anterior cruciate ligament
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Women on estrogen-progestin contraception (Experimental): For women on estrogen-progestin contraception:
  * Correct use of the estrogen-progestin pill in accordance with AMM Or wearing a vaginal ring according to AMM protocol Or wearing a contraceptive skin patch according to AMM protocol
  * Regular cycles of 26 to 33 days
  Interventions: Other: Questionnaire; Other: Beighton test; Other: Lachman Test
- Group 2 Women on progestogen contraception (Experimental): For women on progestin-only contraception:
  o Continuous use of the micro-progestogen or progestogen pill Or subcutaneous hormonal implant, Or a progesterone intrauterine device Or dienogest-type contraception
  Interventions: Other: Questionnaire; Other: Beighton test; Other: Lachman Test
- Group 3 Women without hormonal contraception (Experimental): For women without hormonal contraception :
  * No method of contraception Or copper intrauterine device
  * Regular cycles of 26 to 33 days
  Interventions: Other: Questionnaire; Other: Beighton test; Other: Lachman Test

INTERVENTIONS:
Other: Questionnaire — Questionnaires on contraception and sports activities
Other: Beighton test — A popular screening technique for hypermobility. It consists of a nine-point scale requiring the performance of five maneuvers, four passive bilateral and one active unilateral.
Other: Lachman Test — To perform this test, place your patient in a supine position and bring your patient's test leg to 30 degrees of flexion. Fix the femur with the other hand. Put the tibia in slight external rotation, then try to translate it forwards.
  This test is positive if you feel a soft or limp end or if the anterior part.

SUMMARY:
Women are recognized as being at greater risk of ACL injury, with a risk 6 times higher than that of men. Hyperlaxity is a risk factor for ACL injury, but the pathophysiological basis for this is poorly studied. Hormonal impregnation and certain periods of the menstrual cycle (ovulatory phase) are risk factors for ACL injury. It therefore seems interesting to study the influence of hormonal impregnation on ligament laxity. To date, to our knowledge, no study has investigated such a relationship.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 40 years of age;
* No history of surgery on the 2 lower limbs;
* No change in contraceptive method in the last 6 months;
* Signature of informed consent ;
* Social security affiliation;
* D14 of her menstrual cycle (+/-1 day) (the first day of the cycle (D1) being considered as the first day of menstruation), except for those on unregulated micro-progestogen contraception.

Exclusion Criteria:

* Pregnancy or breastfeeding (check with urine pregnancy test);
* Menopause;
* Surgery: tubal ligation, oophorectomy, adnexectomy, hysterectomy;
* History of inflammatory joint disease, systemic or localized to the knee;
* History of microcrystalline or infectious pathology localized to the knee;
* History of fracture, severe sprain or dislocation of the knee joint;
* History of osteoarticular or congenital diseases that may lead to ACL laxity (e.g. Marfan syndrome, trisomy 21, Ehlers-Danlos syndrome, etc.);
* Signs of hyperlaxity (Beighton test > 4);
* BMI > 25 ;
* Daily alcohol consumption above the thresholds recommended by Public Health in France (more than 2 glasses per day);
* Intense or unusual physical exercise during the last 72 hours before the inclusion visit;
* Inability to understand the protocol;
* Women under guardianship, curatorship or deprived of liberty.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change of anterior tibial translation of the knee with progestin-only hormonal contraception | 24 months
  To show that taking progestin-only hormonal contraception reduces anterior tibial translation of the knee compared with other types of contraception. Anterior tibial knee translation will be considered representative of anterior knee laxity in women on hormonal contraception, using the 30° Lachman test measured with a Lachmeter® digital arthrometer (bilateral examination repeated 3 times on each knee).
  The degree of laxity is assessed using the international IKDC classification:
  * Grade A 0 to 2 mm = normal
  * Grade B 3 to 5 mm = almost normal
  * Grade C 6 to 10 mm = abnormal
  * Grade D > 10 mm = severely abnormal

SECONDARY OUTCOMES:
Change of anterior tibial translation of the knee with progestin-only hormonal contraception or estrogen-only contraception. | 24 months
  To show that taking progestin-only or estrogen-only contraception reduces anterior tibial translation of the knee compared with not taking hormonal contraception. Anterior tibial knee translation will be considered representative of anterior knee laxity in women on hormonal contraception, using the 30° Lachman test measured with a Lachmeter® digital arthrometer (bilateral examination repeated 3 times on each knee).
  The degree of laxity is assessed using the international IKDC classification:
  * Grade A 0 to 2 mm = normal
  * Grade B 3 to 5 mm = almost normal
  * Grade C 6 to 10 mm = abnormal
  * Grade D > 10 mm = severely abnormal
Anterior knee laxity at D14 and D25 of the cycle | 14 or 25 days
  Compare anterior tibial knee translation measured at D14 of the menstrual cycle with that measured at D25 of the menstrual cycle. Anterior tibial knee translation will be considered representative of anterior knee laxity in women on hormonal contraception, using the 30° Lachman test measured with a Lachmeter® digital arthrometer (bilateral examination repeated 3 times on each knee).
  The degree of laxity is assessed using the international IKDC classification:
  * Grade A 0 to 2 mm = normal
  * Grade B 3 to 5 mm = almost normal
  * Grade C 6 to 10 mm = abnormal
  * Grade D > 10 mm = severely abnormal
Variable of height influencing anterior tibial knee translation | 24 months
  Independent factors of ligament laxity in study women (height in meters) will be requested or measured during V1 of the study.
Variable of weight influencing anterior tibial knee translation | 24 months
  Independent factors of ligament laxity in study women (weight in kilograms) will be requested or measured during V1 of the study.
Variable of age influencing anterior tibial knee translation | 24 months
  Independent factors of ligament laxity in study women (age in years) will be requested or measured during V1 of the study.
Variable of duration of contraceptive use influencing anterior tibial knee translation | 24 months
  Independent factors of ligament laxity in study women (duration of contraceptive use in days) will be requested or measured during V1 of the study.
Variable of cycle lenght influencing anterior tibial knee translation | 24 months
  Independent factors of ligament laxity in study women (cycle length in days) will be requested or measured during V1 of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice - Hôpital de l'Archet 2, Nice, Alpes-Maritimes, France